CLINICAL TRIAL: NCT04970901
Title: A Phase 1b Open-Label Study to Evaluate the Safety and Anti-cancer Activity of Loncastuximab Tesirine in Combination With Other Anti-cancer Agents in Patients With Relapsed or Refractory B-cell Non-Hodgkin Lymphoma (LOTIS-7)
Brief Title: A Study to Evaluate the Safety and Anti-cancer Activity of Loncastuximab Tesirine in Combination With Other Anti-cancer Agents in Participants With Relapsed or Refractory B-cell Non-Hodgkin Lymphoma (LOTIS-7)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ADC Therapeutics S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ADCT-402-105; 2021-001071-16 (EudraCT Number)
Record Dates: First submitted 2021-07-12; First posted 2021-07-21 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-06

CONDITIONS: B-Cell Non-Hodgkin Lymphoma; Relapsed B-Cell Non-Hodgkin Lymphoma; Refractory B-Cell Non-Hodgkin Lymphoma
Keywords: B-Cell Non-Hodgkin Lymphoma; Relapsed B-Cell Non-Hodgkin Lymphoma; Refractory B-Cell Non-Hodgkin Lymphoma; Loncastuximab Tesirine
MeSH Terms: conditions — Lymphoma, B-Cell | interventions — loncastuximab tesirine; polatuzumab vedotin; glofitamab; obinutuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part 1 (Dose Escalation): Loncastuximab Tesirine + Polatuzumab Vedotin (Arm C) (Experimental): Participants will receive escalating doses (90 µg/kg to 150 µg/kg) of loncastuximab tesirine on Day (D) 1 of each cycle (where each cycle is 21 days).
  Participants will also receive polatuzumab vedotin at a dose of 1.8 mg/kg on D1 of each cycle, infusion will be started one hour after end of loncastuximab tesirine infusion.
  Interventions: Drug: Loncastuximab Tesirine; Drug: Polatuzumab Vedotin
- Part 1 (Dose Escalation): Loncastuximab Tesirine + Glofitamab (Arm E) (Experimental): Participants will receive escalating doses (90 µg/kg to 150 µg/kg) of loncastuximab tesirine on D2 of Cycle (C) 1 and then D1 of all other cycles (where each cycle is 21 days).
  Participants will also receive glofitamab 2.5 mg on C1 D8, 10 mg on C1 D15 and 30 mg for cycles 2-12 D1.
  In addition participants will receive obinutuzumab pre-treatment 1000 mg on C1 D1.
  Interventions: Drug: Loncastuximab Tesirine; Drug: Glofitamab; Drug: Obinutuzumab
- Part 1 (Dose Escalation): Loncastuximab Tesirine + Mosunetuzumab (Arm F) (Experimental): Participants will receive escalating doses (90 µg/kg to 150 µg/kg) of loncastuximab tesirine on Day (D) 1 of each cycle (where each cycle is 21 days).
  Participants will also receive mosunetuzumab 5 mg on C1 D1, 45 mg for C1 D8, C1 D15 and cycles 2-8 D1.
  Interventions: Drug: Loncastuximab Tesirine; Drug: Mosunetuzumab
- Part 2 (Dose Expansion): Loncastuximab Tesirine + Polatuzumab Vedotin (Arm C) (Experimental): Participants with B-NHL will receive loncastuximab tesirine in combination with polatuzumab vedotin at the maximum tolerated dose (MTD) and/or recommended dose for expansion (RDE) if favorable results of Part 1 are received.
  Interventions: Drug: Loncastuximab Tesirine; Drug: Polatuzumab Vedotin
- Part 2 (Dose Expansion): Loncastuximab Tesirine + Glofitamab (Arm E) (Experimental): Participants with B-NHL will receive loncastuximab tesirine in combination with glofitamab at the MTD and/or RDE if favorable results of Part 1 are received. In addition participants will receive obinutuzumab pre-treatment 1000 mg on C1 D1.
  Interventions: Drug: Loncastuximab Tesirine; Drug: Glofitamab; Drug: Obinutuzumab
- Part 2 (Dose Expansion): Loncastuximab Tesirine + Mosunetuzumab (Arm F) (Experimental): Participants with B-NHL will receive loncastuximab tesirine in combination with mosunetuzumab at the MTD and/or RDE if favorable results of Part 1 are received.
  Interventions: Drug: Loncastuximab Tesirine; Drug: Mosunetuzumab

INTERVENTIONS:
Drug: Loncastuximab Tesirine — Intravenous (IV) infusion
  Other Names: ZYNLONTA; ADCT-402
Drug: Polatuzumab Vedotin — IV infusion
  Arms: Part 1 (Dose Escalation): Loncastuximab Tesirine + Polatuzumab Vedotin (Arm C); Part 2 (Dose Expansion): Loncastuximab Tesirine + Polatuzumab Vedotin (Arm C)
Drug: Glofitamab — IV infusion
  Arms: Part 1 (Dose Escalation): Loncastuximab Tesirine + Glofitamab (Arm E); Part 2 (Dose Expansion): Loncastuximab Tesirine + Glofitamab (Arm E)
Drug: Mosunetuzumab — Subcutaneous (SC) injection
  Arms: Part 1 (Dose Escalation): Loncastuximab Tesirine + Mosunetuzumab (Arm F); Part 2 (Dose Expansion): Loncastuximab Tesirine + Mosunetuzumab (Arm F)
Drug: Obinutuzumab — IV infusion
  Arms: Part 1 (Dose Escalation): Loncastuximab Tesirine + Glofitamab (Arm E); Part 2 (Dose Expansion): Loncastuximab Tesirine + Glofitamab (Arm E)

SUMMARY:
The primary objective of this study is to characterize the safety and tolerability of loncastuximab tesirine in combination with polatuzumab vedotin, glofitamab, or mosunetuzumab, and to identify the maximum tolerated dose (MTD) and/or recommended dose for expansion (RDE) for the combinations.

DETAILED DESCRIPTION:
This is a Phase 1b, multi-center, open-label, multi-arm study to evaluate the safety and anti-cancer activity of loncastuximab tesirine in combination with polatuzumab vedotin, glofitamab, or mosunetuzumab in participants with relapsed or refractory B-cell Non-Hodgkin Lymphoma (R/R B-NHL). The study will enroll approximately 200 participants.

Loncastuximab tesirine (ADCT-402; Zynlonta) is an antibody drug conjugate (ADC), composed of a humanized monoclonal antibody directed against human cluster of differentiation 19 (CD19) conjugated through a cathepsin-cleavable linker to a pyrrolobenzodiazepine (PBD) dimer cytotoxin. Loncastuximab tesirine has been granted by Food and Drug Administration (FDA) as accelerated approval for adult participants with relapsed or refractory large B-cell lymphoma after two or more lines of systemic therapy, including diffuse large B-cell lymphoma (DLBCL) not otherwise specified, DLBCL arising from low grade lymphoma, and high-grade B-cell lymphoma (HGBCL). In the European Union (EU), the European Commission (EC) granted conditional approval for the treatment of adult patients with relapsed or refractory DLBCL and HGBCL, after two or more lines of systemic therapy.

The study includes multiple arms in two parts, Dose Escalation part (Part 1) and Dose Expansion part (Part 2). In Part 1, for the arm of loncastuximab tesirine in combination with polatuzumab vedotin includes DLBCL, HGBCL, follicular lymphoma (FL), mantle cell lymphoma (MCL), marginal zone lymphoma (MZL), and Burkitt lymphoma (BL); for the arms of loncastuximab tesirine in combination with glofitamab or mosunetuzumab include DLBCL, HGBCL, FL, and MZL. In Part 2, participants will be treated at the dose level(s) determined from Part 1. The Sponsor will conduct the safety monitoring and the overall supervision of the study in consultation with the Dose-Escalation Steering Committee (DESC)/Data Safety Monitoring Committee (DSMC).

For each participant, the study will include a Screening Period (of up to 28 days), a Treatment Period (cycles of 21 days), and a Follow-up Period (approximately every 12 week visits for up to two years for Arm C and three years for Arms E and F). Participants may continue treatment for up to one year or until disease progression, unacceptable toxicity, or other discontinuation criteria, whichever occurs first.

Treatment with gemcitabine (Arm A), lenalidomide (Arm B), and umbralisib (Arm D) were removed.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participant aged 18 years or older
* Pathologic diagnosis of relapsed (disease that has recurred following a response) or refractory (disease that failed to respond to prior therapy) B-NHL (2016 World Health Organization classification) who have failed, or been intolerant to any approved therapy and had received at least two systemic treatment regimens in Part 1; and at least one systemic treatment regimen in Part 2

  * LBCL:

Part 2 Arm E enrollment focused on LBCL only

* DLBCL, not otherwise specified (NOS)
* Germinal Center B-cell type
* Activated B-cell type
* Transformed FL (note: patients with transformed FL must have received at least one line of systemic therapy post-transformation to be eligible)
* HGBCL, with MYC and BCL2 and/or BCL6 rearrangements
* HGBCL, NOS
* FL Grade 3b

  * Arm F and Part 1 Arm E:
* All LBCL histologies listed above
* FL (Grade 1-3a)
* MZL

  * For Arm C only:
* All histologies listed above
* DLBCL (including transformed diseases)
* MCL
* BL

  * Life expectancy of at least 24 weeks according to Investigator's judgement
  * Need of systemic treatment for any of the listed indications as assessed by the investigator, including indolent B-NHLs (e.g. FL and MZL)
  * Measurable disease as defined by the 2014 Lugano Classification
  * Availability of formalin-fixed paraffin-embedded tumor tissue block
  * ECOG performance status 0 to 2
  * Adequate organ function
  * Women of childbearing potential (WOCBP) must agree to use a highly effective method of contraception from the time of giving informed consent until at least 10 months after the last dose of loncastuximab tesirine. Men with female partners who are of childbearing potential must agree to use a condom when sexually active or practice total abstinence from the time of giving informed consent the first dose until at least 7 months after the last dose of loncastuximab tesirine. Men must refrain from donating sperm during this same period. Arm E: WOCBP must agree to use contraceptive methods that result in a failure of less than 1% per year or remain abstinent (refrain from heterosexual intercourse) during the treatment period and for at least 18 months after pretreatment with obinutuzumab. Arm F: WOCBP must agree to use contraceptive methods that result in a failure of less than 1% per year or remain abstinent (refrain from heterosexual intercourse) during the treatment period and for at least 3 months after the final dose of mosunetuzumab and tocilizumab (if applicable)
  * Patients 80 years of age and older at the time of signing the informed consent must be deemed fit by Cumulative Illness Rating Scale - Geriatric (CIRS-G scale), defined as no score of 3-4 in any category AND < 5 categories with a score of 2 excluding hematologic criteria

Exclusion Criteria:

* Known history of hypersensitivity resulting in treatment discontinuation to or positive serum human ADA to a CD19 antibody
* Previous therapy with loncastuximab tesirine
* Previous treatment with polatuzumab vedotin, glofitamab or mosunetuzumab (applied to relevant arm and/or cohort of the specific drug administered)

  * Participants who received previous treatment of polatuzumab vedotin containing regimen will be excluded from Arm C
  * Participants who received previous treatment of glofitamab containing regimen will be excluded from Arm E
  * Participants who received previous treatment of mosunetuzumab containing regimen will be excluded from Arm F
* Human immunodeficiency virus (HIV) seropositive
* Serologic evidence of chronic hepatitis B virus (HBV) infection and unable or unwilling to receive standard prophylactic antiviral therapy or with detectable HBV viral load
* Serologic evidence of hepatitis C virus (HCV) infection without completion of curative treatment or with detectable HCV viral load
* History of confirmed progressive multifocal leukoencephalopathy
* History of Stevens-Johnson syndrome, toxic epidermal necrolysis, or macrophage activation syndrome (MAS)/hemophagocytic lymphohistiocytosis (HLH)
* Clinically significant third space fluid accumulation (i.e., ascites requiring drainage or pleural effusion that is either requiring drainage or associated with shortness of breath)
* Breastfeeding or pregnant
* Significant medical comorbidities
* Major surgery, radiotherapy, chemotherapy, or other anti-neoplastic therapy, within 14 days prior to start of study drugs (C1 D1), unless approved by the Sponsor
* Live vaccine within 4 weeks prior to C1D1
* Failure to recover to Grade ≤1 (Common Terminology Criteria for Adverse Events [CTCAE] version 5.0) from acute non-hematologic toxicity (excluding alopecia) due to previous therapy prior to screening
* Active second primary malignancy other than non-melanoma skin cancers, non-metastatic prostate cancer, in situ cervical cancer, ductal or lobular carcinoma in situ of the breast, or other malignancy that the Sponsor's medical monitor and Investigator agree and document should not be exclusionary

Extra Exclusion Criteria for Arms E (includes glofitamab) and F (includes mosunetuzumab) Note: as applicable, the arm-specific exclusion criteria may supersede the general ones, such as stem cell transplant.

* Prior allogeneic stem cell transplant and solid organ transplant
* Autologous stem cell transplant within 100 days prior to C1D1
* History of central nervous system (CNS) lymphoma or leptomeningeal infiltration
* Current or history of CNS disease, such as stroke, epilepsy, CNS vasculitis, or neurodegenerative disease
* Known active infection, reactivation of a latent infection, whether bacterial, viral, fungal, mycobacterial, or other pathogens (excluding fungal infections of nail beds), or any major episode of infection requiring hospitalization or treatment with intravenous (IV) antibiotics within four weeks prior to C1D1
* Active or history of autoimmune disease or immune deficiency, motor neuropathy considered of autoimmune origin and other CNS autoimmune diseases, including but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis, with, with certain exceptions
* Prior treatment with anti-cancer/lymphoma targeted therapies (e.g., tyrosine kinase inhibitors, systemic immunotherapeutic/immunostimulating agents, including, but not limited to, cluster of differentiation 137 agonists or immune checkpoint blockade therapies, including anti-cytotoxic T-lymphocyte-associated antigen 4 (CTLA-4), anti-programmed cell death protein 1 (PD1), and anti-programmed death ligand 1 (PDL1) therapeutic antibodies, radio-immunoconjugates, ADCs, immune/cytokines and monoclonal antibodies) or treatment with systemic immunosuppressive medication (including, but not limited to, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents) within 4 weeks or five half-lives of the drug, whichever is shorter, prior to C1D1, or anticipation of need for systemic immunosuppressive medication during study treatment, with certain exceptions
* Prior treatment with CAR-T-cell therapy within 100 days prior to C1D1; primary refractory patients (progressive or persistent disease within 30 days) to CAR-T-cell therapy are not eligible
* Toxicities from prior anti-cancer therapy including immunotherapy that did not resolve to ≤ Grade 1 with the exception of alopecia, endocrinopathy managed with replacement therapy and stable vitiligo
* Any history of immune-related Grade ≥3 AE with the exception of endocrinopathy managed with replacement therapy
* Ongoing corticosteroid use greater than 25 mg/day of prednisone or equivalent within 4 weeks prior and during study treatment
* Administration of a live attenuated vaccine within 4 weeks prior to the first dose of study treatment or anticipation that such a live attenuated vaccine will be required during the study or within 5 months after last dose of study treatment
* Arm E only: Known history of hypersensitivity to obinutuzumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-06-17 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-10-29 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Experience a Dose-Limiting Toxicity (DLT) | Day 1 to Day 21 of Cycle 1, where a cycle is 21 days
Number of Participants Who Experience a Treatment-emergent Adverse Event (TEAE) | Up to approximately 2 years for Arm C and 3 years for Arms E and F
  Frequency and severity of TEAEs and treatment-emergent serious adverse events (TESAEs). TEAEs and TESAEs will be graded according to Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.
Number of Participants Who Experience an Adverse Event (AE) Leading to Dose Delay | Up to approximately 1 year
Number of Participants Who Experience an Adverse Event (AE) Leading to Dose Interruption | Up to approximately 1 year
Number of Participants Who Experience an Adverse Event (AE) Leading to Dose Reduction | Up to approximately 1 year
Number of Participants Who Experience a Clinically Significant Change from Baseline in Safety Laboratory Measurements | Baseline up to approximately 1 year
Number of Participants Who Experience a Clinically Significant Change from Baseline in Vital Signs | Baseline up to approximately 1 year
Number of Participants Who Experience a Clinically Significant Change from Baseline in Eastern Cooperative Oncology Group (ECOG) Performance Status | Baseline up to approximately 1 year
  ECOG performance status will be measured on a scale from grades 0-5, where a higher grade indicates a worse outcome.
Number of Participants Who Experience a Clinically Significant Change from Baseline in 12-Lead Electrocardiogram (ECG) Measurements | Baseline up to approximately 1 year

SECONDARY OUTCOMES:
Complete Response Rate (CRR) | Up to approximately 2 years for Arm C and 3 years for Arms E and F
Overall Response Rate (ORR) | Up to approximately 2 years for Arm C and 3 years for Arms E and F
Duration of Response (DOR) | Up to approximately 2 years for Arm C and 3 years for Arms E and F
Progression-Free Survival (PFS) | Up to approximately 2 years for Arm C and 3 years for Arms E and F
Relapse-Free Survival (RFS) | Up to approximately 2 years for Arm C and 3 years for Arms E and F
Overall Survival (OS) | Up to approximately 2 years for Arm C and 3 years for Arms E and F
Average Concentration of Loncastuximab Tesirine | Day 1 to end of treatment (up to approximately 1 year)
Maximum Concentration (Cmax) of Loncastuximab Tesirine | Day 1 to end of treatment (up to approximately 1 year)
Time to Maximum Concentration (Tmax) of Loncastuximab Tesirine | Day 1 to end of treatment (up to approximately 1 year)
Area Under the Concentration-Time Curve from Time Zero to the Last Quantifiable Concentration (AUClast) of Loncastuximab Tesirine | Day 1 to end of treatment (up to approximately 1 year)
Area Under the Concentration-Time Curve from Time Zero to the End of the Dosing Interval (AUCtau) of Loncastuximab Tesirine | Day 1 to end of treatment (up to approximately 1 year)
Area Under the Concentration-Time Curve from Time Zero to Infinity (AUCinf) of Loncastuximab Tesirine | Day 1 to end of treatment (up to approximately 1 year)
Apparent Terminal Elimination Half-Life (Thalf) of Loncastuximab Tesirine | Day 1 to end of treatment (up to approximately 1 year)
Apparent Clearance (CL) of Loncastuximab Tesirine | Day 1 to end of treatment (up to approximately 1 year)
Apparent Steady-State Volume of Distribution (Vss) of Loncastuximab Tesirine | Day 1 to end of treatment (up to approximately 1 year)
Accumulation Index (AI) of Loncastuximab Tesirine | Day 1 to end of treatment (up to approximately 1 year)
Number of Participants With Anti-Drug Antibody (ADA) Titers to Loncastuximab Tesirine | Day 1 to end of treatment (up to approximately 1 year)
Arm E Only: Number of Participants With ADA Titers to Glofitamab | Day 1 to end of treatment (up to approximately 1 year)
Arm F Only: Number of Participants With ADA Titers to Mosunetuzumab | Day 1 to end of treatment (up to approximately 1 year)

CONTACTS AND LOCATIONS:
Locations (42):
- United States (25):
  - University of California San Francisco - Fresno Center for Medical Education and Research, Clovis, California
  - Scripps Health - Prebys Cancer Center, San Diego, California
  - Sylvester Comprehensive Cancer Center, Miami, Florida
  - Miami Cancer Institute, Miami, Florida
  - Memorial Cancer Institute - Memorial Hospital West, Pembroke Pines, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - The Blood and Marrow Transplant Group of Georgia, Atlanta, Georgia
  - Mission Cancer + Blood - Mission Cancer Foundation, Des Moines, Iowa
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Columbia University Irving Medical Center, New York, New York
  - Cleveland Clinic Main Campus, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Penn Medicine - Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Allegheny Health Network - West Penn Hospital, Pittsburgh, Pennsylvania
  - Brown University Health - Rhode Island Hospital, Providence, Rhode Island
  - Hollings Cancer Center, Charleston, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Greco-Hainsworth Tennessee Oncology Centers for Research (GHCR), Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Emily Couric Clinical Cancer Center, Charlottesville, Virginia
  - NEXT Virginia (Virginia Cancer Specialists), Fairfax, Virginia
  - Froedtert & Medical College of Wisconsin, Milwaukee, Wisconsin
- Belgium (2):
  - Universitair Ziekenhuis Gent, Ghent
  - Centre Hospitalier Universitaire Universite Catholique de Louvain - Site Godinne, Yvoir
- Czechia (4):
  - Fakultni Nemocnice Brno, Brno, South Moravian
  - Fakultni nemocnice Ostrava, Ostrava
  - Fakultní Nemocnice Královské Vinohrady, Prague
  - Fakultni nemocnice v Motole, Prague
- Italy (4):
  - Azienda Socio Sanitaria Territoriale (ASST) Papa Giovanni XXIII, Bergamo
  - Centro di Ricerche Cliniche - IRCCS Azienda Ospedaliero Universitaria di Bologna, Bologna
  - Azienda Socio Sanitaria Territoriale (ASST) degli Spedali Civili di Brescia, Brescia
  - Istituto Europeo di Oncologia, Milan
- Spain (5):
  - Institut Català d'Oncologia - Hospital Duran i Reynals (ICO L'Hospitalet), Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Complejo Asistencial Universitario de Salamanca - Hospital Clínico, Salamanca
  - Hospital Universitari i Politècnic La Fe, Valencia
- United Kingdom (2):
  - University College London Hospitals NHS Foundation Trust, London
  - Oxford University Hospitals NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: No